CLINICAL TRIAL: NCT04074616
Title: Reducing Anticholinergic Bladder Medication Use in Spinal Cord Injury With Home Neuromodulation
Acronym: TTNS-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Argyrios Stampas, MD, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-19-0518; KL2TR003168 (NIH)
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Chronic Spinal Cord Injury; Neurogenic Bladder
Keywords: electric stimulation
MeSH Terms: conditions — Urinary Bladder, Neurogenic

STUDY DESIGN:
Intervention Model Description: randomized sham-control trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The Study is designed to look at the difference in "high dose" group, which will be submotor amperage, compared to "low dose" which will be set to 1 mA. Both groups will need to stimulate the tibial nerve and visualize toe movement, and then decrease to the amperage of either "high dose" or "low dose." Both groups will use the device for 30 minutes, 5 days per week. A urodynamic study will be performed to measure bladder capacity, sensations while filling, and detrusor pressures before starting using the device and one last time at the end of the study.
  We are also conducting surveys to describe differences in preferences with using bladder medications versus devices.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- High Dose (Experimental)
  Interventions: Device: High Dose
- Control (Other): Low dose TTNS
  Interventions: Device: Low dose

INTERVENTIONS:
Device: High Dose — Electrodes 2 inch by 2 inch will be placed according to anatomic landmarks,with the negative electrode behind the internal malleolus and the positive electrode 10cm superior to the negative electrode, verified with rhythmic flexion of the toes secondary to stimulation of the flexor digitorum and hallicus brevis. The intensity level will be set to the amperage immediately under the threshold for motor contraction. If the patient perceives pain, the intensity will be lowered until comfortable. Stimulation frequency of 10 Hz and pulse width of 200ms in continuous mode will be used.
  Other Names: TTNS stimulation
  Arms: High Dose
Device: Low dose — Toe flexion will be attempted, as in the TTNS protocol. Then the stimulation will be reduced to 1 mA for 30 minutes
  Other Names: TTNS stimulation
  Arms: Control

SUMMARY:
The purpose of this study is to determine the efficacy of home transcutaneous tibial nerve stimulation (TTNS) in spinal cord injury(SCI) and to determine the impact on quality of life using TTNS at home

ELIGIBILITY:
Inclusion Criteria:

* Traumatic and non-traumatic SCI performing IC
* Up to 2 anticholinergic overactive bladder (OAB) medications
* No changes in OAB medications
* Neurologic level of injury above T10
* English and Spanish speaking

Exclusion Criteria:

* Past history of genitourinary diagnoses or surgeries
* History of central nervous system (CNS) disorders and/or peripheral neuropathy
* Pregnancy
* Lower motor neuron bladder
* Concern for tibial nerve pathway injury
* Absence of toe flexion or AD with electric stimulation
* Bladder chemodenervation in past 6 months
* Potential for progressive SCI including neurodegenerative SCI, ALS, cancer myelopathy, Multiple sclerosis, transverse myelitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Argyos Stampas, MD, Principal Investigator — UTHealth
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ackery A, Tator C, Krassioukov A. A global perspective on spinal cord injury epidemiology. J Neurotrauma. 2004 Oct;21(10):1355-70. doi: 10.1089/neu.2004.21.1355. PMID 15672627
- [Background] Weld KJ, Dmochowski RR. Association of level of injury and bladder behavior in patients with post-traumatic spinal cord injury. Urology. 2000 Apr;55(4):490-4. doi: 10.1016/s0090-4295(99)00553-1. PMID 10736489
- [Background] Stohrer M, Blok B, Castro-Diaz D, Chartier-Kastler E, Del Popolo G, Kramer G, Pannek J, Radziszewski P, Wyndaele JJ. EAU guidelines on neurogenic lower urinary tract dysfunction. Eur Urol. 2009 Jul;56(1):81-8. doi: 10.1016/j.eururo.2009.04.028. Epub 2009 Apr 21. PMID 19403235
- [Background] Anderson KD. Targeting recovery: priorities of the spinal cord-injured population. J Neurotrauma. 2004 Oct;21(10):1371-83. doi: 10.1089/neu.2004.21.1371. PMID 15672628
- [Background] Chaabane W, Guillotreau J, Castel-Lacanal E, Abu-Anz S, De Boissezon X, Malavaud B, Marque P, Sarramon JP, Rischmann P, Game X. Sacral neuromodulation for treating neurogenic bladder dysfunction: clinical and urodynamic study. Neurourol Urodyn. 2011 Apr;30(4):547-50. doi: 10.1002/nau.21009. PMID 21488095
- [Background] Chen G, Liao L, Li Y. The possible role of percutaneous tibial nerve stimulation using adhesive skin surface electrodes in patients with neurogenic detrusor overactivity secondary to spinal cord injury. Int Urol Nephrol. 2015 Mar;47(3):451-5. doi: 10.1007/s11255-015-0911-6. Epub 2015 Jan 22. PMID 25609546
- [Background] McDonald JW 3rd, Sadowsky CL, Stampas A. The changing field of rehabilitation: optimizing spontaneous regeneration and functional recovery. Handb Clin Neurol. 2012;109:317-36. doi: 10.1016/B978-0-444-52137-8.00020-6. PMID 23098722
- [Background] Stampas A, Tansey KE. Spinal cord injury medicine and rehabilitation. Semin Neurol. 2014 Nov;34(5):524-33. doi: 10.1055/s-0034-1396006. Epub 2014 Dec 17. PMID 25520024
- [Background] Stampas A, York HS, O'Dell MW. Is the Routine Use of a Functional Electrical Stimulation Cycle for Lower Limb Movement Standard of Care for Acute Spinal Cord Injury Rehabilitation? PM R. 2017 May;9(5):521-528. doi: 10.1016/j.pmrj.2017.03.005. No abstract available. PMID 28526124
- [Background] Stampas A, Korupolu R, Zhu L, Smith CP, Gustafson K. Safety, Feasibility, and Efficacy of Transcutaneous Tibial Nerve Stimulation in Acute Spinal Cord Injury Neurogenic Bladder: A Randomized Control Pilot Trial. Neuromodulation. 2019 Aug;22(6):716-722. doi: 10.1111/ner.12855. Epub 2018 Oct 3. PMID 30284350
- [Background] del Popolo G, Mencarini M, Nelli F, Lazzeri M. Controversy over the pharmacological treatments of storage symptoms in spinal cord injury patients: a literature overview. Spinal Cord. 2012 Jan;50(1):8-13. doi: 10.1038/sc.2011.110. Epub 2011 Nov 1. PMID 22042300
- [Background] Canbaz Kabay S, Kabay S, Mestan E, Cetiner M, Ayas S, Sevim M, Ozden H, Karaman HO. Long term sustained therapeutic effects of percutaneous posterior tibial nerve stimulation treatment of neurogenic overactive bladder in multiple sclerosis patients: 12-months results. Neurourol Urodyn. 2017 Jan;36(1):104-110. doi: 10.1002/nau.22868. Epub 2015 Sep 9. PMID 26352904
- [Background] Sirls ER, Killinger KA, Boura JA, Peters KM. Percutaneous Tibial Nerve Stimulation in the Office Setting: Real-world Experience of Over 100 Patients. Urology. 2018 Mar;113:34-39. doi: 10.1016/j.urology.2017.11.026. Epub 2017 Nov 28. PMID 29196071
- [Background] Fougere RJ, Currie KD, Nigro MK, Stothers L, Rapoport D, Krassioukov AV. Reduction in Bladder-Related Autonomic Dysreflexia after OnabotulinumtoxinA Treatment in Spinal Cord Injury. J Neurotrauma. 2016 Sep 15;33(18):1651-7. doi: 10.1089/neu.2015.4278. Epub 2016 Apr 13. PMID 26980078
- [Background] Sievert KD, Amend B, Gakis G, Toomey P, Badke A, Kaps HP, Stenzl A. Early sacral neuromodulation prevents urinary incontinence after complete spinal cord injury. Ann Neurol. 2010 Jan;67(1):74-84. doi: 10.1002/ana.21814. PMID 20186953
- [Background] de Seze M, Raibaut P, Gallien P, Even-Schneider A, Denys P, Bonniaud V, Game X, Amarenco G. Transcutaneous posterior tibial nerve stimulation for treatment of the overactive bladder syndrome in multiple sclerosis: results of a multicenter prospective study. Neurourol Urodyn. 2011 Mar;30(3):306-11. doi: 10.1002/nau.20958. Epub 2011 Feb 8. PMID 21305588
- [Background] Sanford MT, Suskind AM. Neuromodulation in neurogenic bladder. Transl Androl Urol. 2016 Feb;5(1):117-26. doi: 10.3978/j.issn.2223-4683.2015.12.01. PMID 26904417
- [Background] Stampas A, Gustafson K, Korupolu R, Smith C, Zhu L, Li S. Bladder Neuromodulation in Acute Spinal Cord Injury via Transcutaneous Tibial Nerve Stimulation: Cystometrogram and Autonomic Nervous System Evidence From a Randomized Control Pilot Trial. Front Neurosci. 2019 Feb 19;13:119. doi: 10.3389/fnins.2019.00119. eCollection 2019. PMID 30837835
- [Background] Dubeau CE. The aging lower urinary tract. J Urol. 2006 Mar;175(3 Pt 2):S11-5. doi: 10.1016/S0022-5347(05)00311-3. PMID 16458733
- [Background] Schurch B, Denys P, Kozma CM, Reese PR, Slaton T, Barron R. Reliability and validity of the Incontinence Quality of Life questionnaire in patients with neurogenic urinary incontinence. Arch Phys Med Rehabil. 2007 May;88(5):646-52. doi: 10.1016/j.apmr.2007.02.009. PMID 17466735
- [Background] Welk B, Lenherr S, Elliott S, Stoffel J, Presson AP, Zhang C, Myers JB. The Neurogenic Bladder Symptom Score (NBSS): a secondary assessment of its validity, reliability among people with a spinal cord injury. Spinal Cord. 2018 Mar;56(3):259-264. doi: 10.1038/s41393-017-0028-0. Epub 2017 Nov 29. PMID 29184133
- [Background] Welk B, Carlson K, Baverstock R. A pilot study of the responsiveness of the Neurogenic Bladder Symptom Score (NBSS). Can Urol Assoc J. 2017 Dec;11(12):376-378. doi: 10.5489/cuaj.4833. Epub 2017 Nov 1. No abstract available. PMID 29257742
- [Background] Ibrahim JG, Molenberghs G. Missing data methods in longitudinal studies: a review. Test (Madr). 2009 May 1;18(1):1-43. doi: 10.1007/s11749-009-0138-x. PMID 21218187
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Background] Morisky DE, Ang A, Krousel-Wood M, Ward HJ. Predictive validity of a medication adherence measure in an outpatient setting. J Clin Hypertens (Greenwich). 2008 May;10(5):348-54. doi: 10.1111/j.1751-7176.2008.07572.x. PMID 18453793
- [Background] Walsh JC, Mandalia S, Gazzard BG. Responses to a 1 month self-report on adherence to antiretroviral therapy are consistent with electronic data and virological treatment outcome. AIDS. 2002 Jan 25;16(2):269-77. doi: 10.1097/00002030-200201250-00017. PMID 11807312
- [Background] Gruber-Baldini AL, Velozo C, Romero S, Shulman LM. Validation of the PROMIS(R) measures of self-efficacy for managing chronic conditions. Qual Life Res. 2017 Jul;26(7):1915-1924. doi: 10.1007/s11136-017-1527-3. Epub 2017 Feb 26. PMID 28239781

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Dose | Control
Started | 25 | 25
Completed | 20 | 22
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose | Control | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [29 to 49] | 41 [32 to 48] | 38 [30 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 22 | 21 | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
Number of Participants with Tetraplegia [Count of Participants; unit: Participants] | 13 | 10 | 23
Number of Participants with imaging pathology [Count of Participants; unit: Participants] — Population: 9 participants in the high dose arm did not receive Bladder and Kidney imaging. 11 participants in the control arm did not receive Bladder and Kidney imaging.
  Participants
    Hydronephrosis: number analyzed (Participants) | 16 | 14 | 30
    Hydronephrosis | 0 | 0 | 0
    Nephrolithiasis: number analyzed (Participants) | 16 | 14 | 30
    Nephrolithiasis | 3 | 1 | 4
    Bladder stones: number analyzed (Participants) | 16 | 14 | 30
    Bladder stones | 1 | 0 | 1
    Hydroureter: number analyzed (Participants) | 16 | 14 | 30
    Hydroureter | 1 | 0 | 1
Number of Participants with Bladder and Kidney Imaging [Count of Participants; unit: Participants] | 16 | 14 | 30
Years from injury to cystometrogram [Median (Inter-Quartile Range); unit: years] — Population: Data were not collected from participant in the high dose arm.
  years
    number analyzed (Participants) | 24 | 25 | 49
    (all) | 10.8 [6.9 to 20.3] | 8.9 [2.9 to 16.6] | 10.3 [4.5 to 19.9]
Number of Overactive Bladder medications [Mean (Standard Deviation); unit: medications] | 1.4 (0.5) | 1.2 (0.4) | 1.3 (0.5)
Creatinine [Mean (Standard Deviation); unit: milligrams per decilitre] — Population: Data were not collected for 18 participants in the high does arm. Data were not collected for 14 participants in the control arm.
  milligrams per decilitre
    number analyzed (Participants) | 7 | 11 | 18
    (all) | .85 (.23) | .68 (.19) | .74 (.21)
Asia Impairment Scale Classification [Count of Participants; unit: Participants] — The Asia Impairment Scale (AIS) categorizes spinal cord injury severity based on sensory and motor function loss.
  AIS Classification:
  A = Complete: No motor/sensory function in the sacral segments S4-S5
  B = Incomplete: Sensory but not motor function below the neurological level, includes the sacral segments S4-S5
  C = Incomplete: Below the neurological level, motor function preserved and more than 50% of key muscles have a muscle grade < 3
  D = Incomplete: Below the neurological level, motor function persevered and at least 50% of key muscles have a muscle grade ≥3
  Participants
    A | 14 | 14 | 28
    B | 6 | 2 | 8
    C | 4 | 4 | 8
    D | 1 | 5 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reduction in Bladder Medication
Time Frame: baseline, 3 months
Population: Data were not collected for 5 participants in the high dose arm. Data were not collected for 3 participants in the control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose | Control
Number analyzed (Participants) | 20 | 22
Participants | 19 | 15

2. Primary Outcome: Number of Participants With a Change in Neurogenic Bladder Symptom Score (NBSS) Scale From Baseline
Description: The Neurogenic Bladder Symptom (NBSS) Score is a questionnaire that measures bladder symptoms, with total score ranging from 0 to 74; a higher score indicating a worse outcome.
  Scores at baseline are compared to scores at 3 months, and a change is reported categorically as follows:
  Stable: A score change within + 5 or -5 points (not including 5)
  Worse: A score increase of 5 points or more from baseline
  Improved: A score decrease of 5 points or more from baseline
  These categories are mutually exclusive and exhaustive; each participant will fit into only one category based on their score change
Time Frame: Baseline, 3 months
Population: Data were not collected for 9 participants in the high dose arm. Data were not collected for 4 participants in the control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose | Control
Number analyzed (Participants) | 16 | 21
Participants
  Stable | 8 | 7
  Improved | 7 | 11
  Worse | 1 | 3

3. Primary Outcome: Number of Participants With Reduced Neurogenic Bladder Symptoms (NGB) as Measured by the Voiding Diary
Time Frame: baseline, 3 months
Population: Data were not collected from 11 participants in the high dose arm. Data were not collected for 7 participants in the control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose | Control
Number analyzed (Participants) | 14 | 18
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With a Change in the Incontinence Quality of Life Questionnaire Score From Baseline
Description: The Incontinence Quality of Life questionnaire assesses the impact of urinary incontinence on a person's quality of life. The total score ranges from 0 to 100, a lower score indicating a worse outcome. Scores at baseline are compared to scores at 3 months, and a change is reported as categorically as follows:
  Stable: A score change within +4 or -4 points (not including 4)
  Worse: A score decrease of 4 or more points from baseline
  Improved: A score increase of 4 or more points from baseline
  These categories are mutually exclusive and exhaustive; each participant will fit into only one category based on their score change.
Time Frame: baseline, 3 months
Population: Data were not collected for 8 participants in the high dose arm. Data were not collected for 4 participants in the control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose | Control
Number analyzed (Participants) | 17 | 21
Participants
  stable | 4 | 6
  improved | 6 | 4
  worse | 7 | 11

5. Secondary Outcome: Number of Participants With Decreased Anticholinergic Side Effects as Measured by the Anticholinergic Side Effects Survey
Time Frame: baseline, 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose | Control
Number analyzed (Participants) | 20 | 22
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Increased or Stable Bladder Capacity as Assessed by the Urodynamic Study
Time Frame: baseline, 3 months
Population: Data were not collected for 5 participants in the high dose arm. Data were not collected for 4 participants in the control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose | Control
Number analyzed (Participants) | 20 | 21
Participants | 12 | 14

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | High Dose | Control
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 4/25 | 6/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose (N=25) | Control (N=25)
Urinary Tract Infection (Renal and urinary disorders) | 4 | 6
Pressure injury (Injury, poisoning and procedural complications) | 1 | 0
COVID (General disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
The COVID-19 pandemic imposed constraints on participants' ability to travel and communicate, leading to dropouts, as well as affecting research staffing and the ability to perform research.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT04074616/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT04074616/ICF_001.pdf